CLINICAL TRIAL: NCT05127707
Title: Effect of Exposure to Visual Campaigns and Narrative Vignettes on Addiction Stigma Among Health Professionals: A Randomized Experiment
Brief Title: Strategies to Reduce Addiction Stigma Among Health Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB14743
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Opioid Use Disorder; Substance Use Disorders; Stigma, Social
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- No exposure control group (No Intervention): This group was not exposed to any message frame.
- Words Matter - Visual Campaign (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the importance of use of non-stigmatizing language regarding substance use disorder and opioid use disorder in clinical settings.
  Interventions: Behavioral: Words Matter - Visual Campaign
- Words Matter - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the importance of use of non-stigmatizing language regarding substance use disorder and opioid use disorder in clinical settings and a narrative vignette told from the perspective of a person with opioid use disorder.
  Interventions: Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder) Experimental: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician)
- Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the importance of use of non-stigmatizing language regarding substance use disorder and opioid use disorder in clinical settings and a narrative vignette told from the perspective of a clinician.
  Interventions: Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician)
- Words Matter - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the importance of use of non-stigmatizing language regarding substance use disorder and opioid use disorder in clinical settings and a narrative vignette told from the perspective of a health system administrator/leader.
  Interventions: Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator)
- Medication Treatment Works - Visual Campaign (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the effectiveness of medications for treating opioid use disorder in saving lives.
  Interventions: Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign
- Medication Treatment Works - Visual Campaign & Narrative Vignette (Person with OUD) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the effectiveness of medications for treating opioid use disorder in saving lives and a narrative vignette told from the perspective of a person with opioid use disorder.
  Interventions: Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder)
- Medication Treatment Works - Visual Campaign & Narrative Vignette (Clinician) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the effectiveness of medications for treating opioid use disorder in saving lives and a narrative vignette told from the perspective of a clinician.
  Interventions: Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Clinician)
- Medication Treatment Works - Visual Campaign & Narrative Vignette (Health System Administrator) (Experimental): Participants randomized to this arm were exposed to a visual campaign communicating the effectiveness of medications for treating opioid use disorder in saving lives and a narrative vignette told from the perspective of a health system administrator/leader.
  Interventions: Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator)

INTERVENTIONS:
Behavioral: Words Matter - Visual Campaign — Visual campaign emphasizing the importance of using non-stigmatizing language related to substance use and opioid use disorder in clinical settings.
  Arms: Words Matter - Visual Campaign
Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder) Experimental: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician) — Visual campaign emphasizing the importance of using non-stigmatizing language related to substance use and opioid use disorder in clinical settings combined with a narrative vignette told from the perspective of a person with opioid use disorder
  Arms: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder)
Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician) — Visual campaign emphasizing the importance of using non-stigmatizing language related to substance use and opioid use disorder in clinical settings combined with a narrative vignette told from the perspective of a clinician working with patients with opioid use disorder
  Arms: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Clinician)
Behavioral: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator) — Visual campaign emphasizing the importance of using non-stigmatizing language related to substance use and opioid use disorder in clinical settings combined with a narrative vignette told from the perspective of a health system administrator/leader
  Arms: Words Matter - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator)
Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign — Visual campaign emphasizing the effectiveness and value of medications to treat opioid use disorder in saving lives
  Arms: Medication Treatment Works - Visual Campaign
Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Person with Opioid Use Disorder) — Visual campaign emphasizing the effectiveness and value of medications to treat opioid use disorder in saving lives combined with a narrative vignette told from the perspective of a person with opioid use disorder
  Arms: Medication Treatment Works - Visual Campaign & Narrative Vignette (Person with OUD)
Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Clinician) — Visual campaign emphasizing the effectiveness and value of medications to treat opioid use disorder in saving lives combined with a narrative vignette told from the perspective of a clinician who treats people with opioid use disorder
  Arms: Medication Treatment Works - Visual Campaign & Narrative Vignette (Clinician)
Behavioral: Medication Treatment for Opioid Use Disorder Works - Visual Campaign & Narrative Vignette (Messenger: Health System Administrator) — Visual campaign emphasizing the effectiveness and value of medications to treat opioid use disorder in saving lives combined with a narrative vignette told from the perspective of a health system administrator/leader
  Arms: Medication Treatment Works - Visual Campaign & Narrative Vignette (Health System Administrator)

SUMMARY:
The aim of this study was to evaluate the effects of exposure to stigma reduction message frames communicated by visual campaigns and narrative vignettes among a national sample of health professionals.

DETAILED DESCRIPTION:
This randomized experiment evaluated the impact of exposure to message frames communicating the importance of non-stigmatizing language regarding addiction and the effectiveness of medication treatment for opioid use disorder delivered through a visual campaign alone or through a visual campaign in addition to a narrative vignette from the perspective of one of three messengers (a person with opioid use disorder, a clinician, or a health system leader) on attitudes toward people with opioid use disorder and medications for treating opioid use disorder among a national sample of health professionals.

ELIGIBILITY:
Inclusion Criteria:

* employed as health professional in the United States, including clinicians (e.g., physicians, nurses, physician assistants, pharmacists, and optometrists), technicians and technologists (e.g., laboratory technologist or technician, emergency medical technician, paramedic, licensed practical or licensed vocational nurse, medical records or health information technician, etc.), health aids and assistants (e.g., nursing aide, home health aide, medical assistant, pharmacy aide, phlebotomist, etc.)
* participant in existing web-based survey panel (IPSOS's KnowledgeNetworks panel and partner opt-in panel)

Exclusion Criteria:

* not employed in health profession
* not able to complete experiment and survey in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1842 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Rating of willingness to have person with opioid use disorder marry into their family | Measured immediately post-exposure to message frame intervention
  Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 5 indicating greater unwillingness and 1 indicating greater willingness to have a person with opioid use disorder marry into the family. Measured via survey questionnaire.
Rating of willingness to have person with opioid use disorder as a neighbor | Measured immediately post-exposure to message frame intervention
  Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 5 indicating greater unwillingness and 1 indicating greater willingness to have a person with opioid use disorder as a neighbor. Measured via survey questionnaire.
Rating of agreement that opioid use disorder is a medical condition | Measured immediately post-exposure to message frame intervention
  Rating of agreement with statement "Opioid use disorder is a chronic medical condition like diabetes mellitus" on 5-point Likert scale with 5 indicating strong disagreement and 1 indicating strong agreement. Measured via survey questionnaire.
Rating of agreement that individuals with opioid use disorder are to blame | Measured immediately post-exposure to message frame intervention
  Rating of agreement with statement "Individuals with opioid use disorder only have themselves to blame for their problem" on 5-point Likert scale with 5 indicating strong disagreement and 1 indicating strong agreement. Measured via survey questionnaire.
Rating of support for increasing government spending on opioid use disorder treatment | Measured immediately post-exposure to message frame intervention
  Rating of support for increasing government spending on treatment of opioid use disorder with 5 indicating strongly favoring and 1 indicating strongly opposing. Measured via survey questionnaire.
Feeling thermometer measure of warmth toward people with opioid use disorder | Measured immediately post-exposure to message frame intervention
  Rating of warmth felt toward people with opioid use disorder with 0 indicating extremely cold and 100 indicating extremely warm. Measured via survey questionnaire.

SECONDARY OUTCOMES:
Stigmatizing Language - Addict | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "addict" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - Substance abuse | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "substance abuse" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - dirty | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "'dirty' in reference to the result from a drug test" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - clean | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "'clean' in reference to the result from a drug test" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - addicted baby | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "addicted baby" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - person with substance use disorder | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "person with substance use disorder" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - substance use | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "substance use" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - negative test result | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "negative test result" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - positive test result | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "positive test result" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Stigmatizing Language - baby born with neonatal opioid withdrawal syndrome | Measured immediately post-exposure to message frame intervention
  Rating of agreement that term "baby born with neonatal opioid withdrawal syndrome" appropriate in a clinical care setting with 1 indicating strongly agree (that term is appropriate) and 5 indicating strongly disagree (that term is appropriate). Measured via survey questionnaire.
Willingness to sign pledge committing to using non-stigmatizing language | Measured immediately post-exposure to message frame intervention
  Binary (yes/no) measure of whether participant is willing to sign a pledge committing to using non-stigmatizing language related to substance use disorder in clinical settings. Measured via survey questionnaire.
Perception of opioid use disorder treatment effectiveness | Measured immediately post-exposure to message frame intervention
  Participant perception of whether there is a treatment for opioid use disorder that is effective for a long period of time (three close-ended response options: yes, there is a treatment; no, there isn't such a treatment; don't know). Measured via survey questionnaire.
Rating of willingness to have person taking medication marry into their family | Measured immediately post-exposure to message frame intervention
  Rating of willingness to have person taking medication to treat opioid use disorder marry into family. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 5 indicating greater unwillingness and 1 indicating greater willingness to have a person taking medication to treat opioid use disorder marry into the family. Measured via survey questionnaire.
Rating of willingness to have person taking medication marry as a neighbor | Measured immediately post-exposure to message frame intervention
  Rating of willingness to have person taking medication to treat opioid use disorder as a neighbor. Item from the Social Distance Scale that measures one element of stigma (desire for social distance). Measured on 5-point Likert scale with 5 indicating greater unwillingness and 1 indicating greater willingness to have a person taking medication to treat opioid use disorder as a neighbor. Measured via survey questionnaire.
Rating of strength/weakness of person taking medication | Measured immediately post-exposure to message frame intervention
  Rating of strength/weakness of person taking medication to treat opioid use disorder on 5-point Likert scale with 5 indicating strong and 1 indicating weak. This is a semantic differential measure. Measured via survey questionnaire.
Rating of agreement that recovery is possible | Measured immediately post-exposure to message frame intervention
  Rating of agreement with statement "Most people with opioid use disorder will, with medication treatment, get well and return to productive lives" on a 5-point Likert scale with 5 indicating strongly disagree and 1 indicating strongly agree. Measured via survey questionnaire.
Feeling thermometer measure of warmth toward people taking medication | Measured immediately post-exposure to message frame intervention
  Rating of warmth felt toward people taking medication to treat opioid use disorder with 0 indicating extremely cold and 100 indicating extremely warm. Measured via survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alene Kennedy-Hendricks, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennedy-Hendricks A, McGinty EE, Summers A, Krenn S, Fingerhood MI, Barry CL. Effect of Exposure to Visual Campaigns and Narrative Vignettes on Addiction Stigma Among Health Care Professionals: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2146971. doi: 10.1001/jamanetworkopen.2021.46971. PMID 35119460